CLINICAL TRIAL: NCT02457455
Title: Inflight Emergencies During Eurasian Flights
Brief Title: Urgent Medical and Surgical Conditions During Flights
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Antalya TRH 002
Record Dates: First submitted 2015-05-20; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Syncope; Arrest; Vertigo; Pain; Chronic Obstructive Pulmonary Disease; Hypertension; CAD
Keywords: inflight emergencies
MeSH Terms: conditions — Syncope; Heart Arrest; Vertigo; Pain; Pulmonary Disease, Chronic Obstructive; Hypertension

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sick passangers: Passengers or cabincreew whom needed urgent medical supports during flights with completed medical records. (Aforementioned Flight Company records complaints, symptoms and diagnoses, demographic data, the mortality of those who request medical aid, whether medical treatment is performed by the cabin crew or by a medical professional on the plane, as well as those conditions which resulted in an emergency landing and dead). All ages are included.

SUMMARY:
The aim of this study is to evaluate the incidence and status of urgent medical conditions. After defining the urgent situations, the investigators will evaluate the adequacy of the standard medical kits and trainings.

DETAILED DESCRIPTION:
In this study, the incidence and status of urgent medical conditions, the attitudes of health professionals who encounter such conditions, adequacy of Aerospace Medical Association (ASMA) suggested medical kits and training of cabin crew in data-received-company aircrafts and the demographic data of patients have been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All passengers (no age limitations) needed urgent medical support during flights

Exclusion Criteria:

* Patients whom medical urgency records are insufficient

Ages: 2 Weeks to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All passengers who needs urgent medical support
Sampling Method: Probability Sample
Enrollment: 1312 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of the urgent medical demands during flights | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kesapli, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of Emergency, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Thibeault C, Evans AD. AsMA Medical Guidelines for Air Travel: stresses of flight. Aerosp Med Hum Perform. 2015 May;86(5):486-7. doi: 10.3357/AMHP.4225.2015. PMID 25945668
- [Background] Ruskin KJ. In-flight medical emergencies: time for a registry? Crit Care. 2009;13(1):121. doi: 10.1186/cc7715. Epub 2009 Feb 25. PMID 19291266
- [Background] Ruskin KJ, Hernandez KA, Barash PG. Management of in-flight medical emergencies. Anesthesiology. 2008 Apr;108(4):749-55. doi: 10.1097/ALN.0b013e31816725bc. No abstract available. PMID 18362607
- [Background] Lyznicki JM, Williams MA, Deitchman SD, Howe JP 3rd; Council on Sceientific Affairs, American Medical Association. Inflight medical emergencies. Aviat Space Environ Med. 2000 Aug;71(8):832-8. PMID 10954361